CLINICAL TRIAL: NCT05597813
Title: The Role of Topical Timolol 0.5% in Wound Healing and Scar Improvement Following Atrophic Acne Scar Microneedling
Brief Title: Topical Timolol 0.5% in Atrophic Acne Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: atrophic acne scars
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): microneedling group
  Interventions: Procedure: microneedling
- Group B (Active Comparator): microneedling plus timolol group
  Interventions: Procedure: microneedling with topical timolol 0.5%

INTERVENTIONS:
Procedure: microneedling — 15 patients will be subjected to microneedling alone. Selected patients will receive one session with two weeks interval till complete clearance or up to 6 sessions.
  Arms: Group A
Procedure: microneedling with topical timolol 0.5% — 15 patients will be subjected to microneedling with topical timolol 0.5%.Selected patients will receive one session with two weeks interval till complete clearance or up to 6 sessions.
  Arms: Group B

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of microneedling combined with topical timolol 0.5% in the treatment of atrophic acne scars.

DETAILED DESCRIPTION:
Acne vulgaris (AV) is a common chronic inflammatory disease of skin that develops from sebaceous glands associated with hair follicles. Typically AV begins at puberty and may continue through adulthood affecting the comedogenic areas of face, back and chest (Mazzetti et al., 2019).

One of the undesirable outcomes of acne is acne scars that are divided into two main types based on a loss (atrophic) or gain (hypertrophic) of collagen. Atrophic type is the most common type, further subdivided into three subtypes: icepick, boxcar and rolling scar (Bahl et al., 2020).

Post acne scars occur in nearly 75% of patients with acne affecting both male and female equally (Khunger and Kumar, 2012). Acne scars impair quality of life and may be a risk factor for depression, suicide, low academic performance and unemployment (Sood et al., 2020).

There are different therapeutic modalities for atrophic acne scars including microneedling, chemical peeling, laser, filler, surgical procedures (punch excision, punch grafts) and fat transfer (Pavlidis and Katsambus, 2017).

Microneedling is considered safe for all skin types. It is performed by dermapen or dermaroller to induce new collagen formation that remains for a few months after the procedure (Cohen and Elbuluk, 2016).

Microneedling enhances the effect of topical preparations when used combined with them due to increasing their absorption by creating small channels through the epidermis to the dermis (Jaffe, 1981).

Ghassemi et al. (2021) observed that application of 0.5% timolol after TCA-CROSS caused a slight increase in scar improvement with more physician and patients' satisfaction.

Timolol, a beta-adrenergic receptor blocker, improves healing of skin wounds by increasing the phosphorylation of extracellular signal regulated kinases (ERK) leading to keratinocyte migration (Zeigler et al., 1999). Also, ERK initiate signaling cascades leading to fibroblast mitosis and proliferation with regulation of fibroblast functions in replacement of disorganized collagen and the reposition of the extracellular matrix (de Araújo et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

1. All types of facial atrophic acne scars
2. Patients aged >18 years
3. Both sexes

Exclusion Criteria:

1. Pregnancy and lactation
2. Active acne or any active facial lesion
3. History of keloid scar
4. History of systemic diseases as DM or hypotension
5. Bleeding and coagulation disorders
6. Infection and immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Goodman and Baron's acne scar grading system | through study completion, an average of 9 months
  Grade 1 Erythematous hypo or hyperpigmented flat marks Grade 2 Mild atrophy not obvious at social distance of >/=50 cm or easily covered by makeup or beard hair in male Grade 3 Moderate atrophy obvious at social distance of >/=50 cm, not easily covered by makeup or beard hair but able to be flattened by manual stretching of the skin Grade 4 Sever atrophy obvious at social distance >50 cm, not easily covered by makeup and not able to be flattened by manual stretching of skin
Quartile grading system | through study completion, an average of 9 months
  The improvement of patients is evaluated as follow:
  Poor (improvement < 25%) Mild (improvement 26%-50%) Good (improvement 51%-75%) Excellent (improvement >75%) (Saadawi et al., 2018)
5 point scale for evaluating patient's satisfaction | through study completion, an average of 9 months
  None (no satisfaction) Mild (1%-25% satisfaction) Moderate (26%-50% satisfaction) Good (51%-75% satisfaction) Very good (76%-100% satisfaction) (El Domyati et al., 2015)
Pain assessment | through study completion, an average of 9 months
  Pain during the session will be assessed and graded as mild, moderat and sever (Saadawi et al., 2018).